CLINICAL TRIAL: NCT00403806
Title: Antiemetic and Analgesic Efficacy and Safety of Dexamethasone for Paediatric Adeno-tonsillectomy - A Randomised, Placebo-controlled, Double-blind, Dose-finding Study
Brief Title: Dexamethasone for Paediatric Adeno-tonsillectomy - A Dose-finding Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: drug-related harm
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Christoph Czarnetzki MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAC 04-005; Swissmedic DR 3028
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2009-01

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain
Keywords: Adenotonsillectomy; Pediatrics; Postoperative Nausea and Vomiting; Pain; Oral intake; Dexamethasone; Dose finding
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative; Pain | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Intravenous dexamethasone 0.05 mg per kg bodyweight
  Interventions: Drug: dexamethasone
- 2 (Active Comparator): Intravenous dexamethasone 0.15 mg per kg bodyweight
  Interventions: Drug: Dexamethasone
- 3 (Active Comparator): Intravenous dexamethasone 0.5 mg per kg bodyweight
  Interventions: Drug: dexamethasone
- 4 (Placebo Comparator): Intravenous saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: dexamethasone — intravenous dexamethasone 0.05 mg per kg bodyweight
  Other Names: Mephamesone
  Arms: 1
Drug: Dexamethasone — Intravenous dexamethasone 0.15 mg per kg bodyweight
  Other Names: mephamesone
  Arms: 2
Drug: dexamethasone — Intravenous dexamethasone 0.5 mg per kg bodyweight
  Other Names: mephamesone
  Arms: 3
Drug: Saline — Intravenous saline
  Other Names: mephamesone
  Arms: 4

SUMMARY:
Adeno-tonsillectomy is a commonly performed surgical procedure in children. Main morbidities are postoperative pain, nausea and vomiting, and haemorrhage. Non-steroidal anti-inflammatory drugs (NSAIDs)widely used for paincontrol increase the risk of postoperative bleeding and reoperation. Dexamethasone is an powerful antiemetic and has shown analgesic efficacy. Antiemetic and analgesic dose-response has never been established.

DETAILED DESCRIPTION:
1. Primary objective: To investigate the dose-effect relationship of prophylactic single-dose dexamethasone for the prevention of PONV in children undergoing adeno-tonsillectomy.
2. Secondary objective:To investigate the dose-effect relationship of prophylactic single-dose dexamethasone for the prevention of postoperative pain and its effect on general outcome in children undergoing adeno-tonsillectomy. To investigate the safety of dexamethasone in children undergoing adeno-tonsillectomy.
3. Study Population:Children, aged 3 to 16 years, scheduled for elective tonsillectomy with or without adenoidectomy, and with or without ear tubes will be included. Children will stay the first postoperative night at the hospital and will be discharged the day after surgery.
4. Randomisation and blinding:Children will be randomised to one of four groups of equal size:

   Group 1: Placebo NaCL 0.9%,Group 2:Dexa 0.05 mg/kg, Group 3: Dexa 0.15 mg/kg, Group 4:Dexa 0.5 mg/kg

   Indistinguishable 20 ml ampoules will be prepared and randomised by the Hospital Pharmacy. Children will receive 0.5 ml/kg of the solution as an IV bolus after induction of anaesthesia. The maximum volume of dexamethasone injected will be limited to 20 ml (corresponding to a maximum dose of 20 mg in a child with ≥40 kg bodyweight).

   Standardized Anesthesia technique and surgical procedure
5. Variables measured

5.1. Intraoperatively

* Type of surgery
* Surgical time
* Dose of opioid

5.2. Postoperatively

Follow up will be during the hospital stay, through a telephone interview 48 hours after surgery, and through a surgical control (standard procedure) at about one week. Preoperatively, parents and children will be instructed in the evaluation of pain. Parents will be given a questionnaire to be filled in twice daily (morning and evening) after discharge of the child, and to bring it back to the routine postoperative surgical control at one week (or to send it back by post).

Endpoint PONV

* Cumulative incidence of vomiting (including retching) during the first 6 postoperative hours.
* Cumulative incidence of nausea during the first 6 postoperative hours. Nausea is only recorded if the child is able to express the sensation of nausea.
* Cumulative incidence of vomiting (including retching) during the first 24 postoperative hours.
* Cumulative incidence of nausea during the first 24 postoperative hours. Rescue medication for PONV is with ondansetron (Zofran) 50 µg/kg IV or droperidol 20 µg/kg IV. Rescue antiemesis will be recorded.

Endpoint pain intensity In hospitalised children, pain assessment will be with the revised Faces Pain Scale (FPS-r) [Hicks et al, 2001] and with the conventional 0-10 cm Visual Analogue Scale (VAS). The FPS-r was adapted from the Faces Pain Scale [Bieri et al, 1990] in order to make it possible to score on the widely accepted 0-10 point metric. It shows a close linear relationship with the visual analogue pain scale across the age range from 4 to 16 years. In the case that a younger child is not able to express adequately its pain with the FPS-r or with the VAS we will use the CHEOP Scale (Children of Eastern Ontario Pain Scale); this is a behavioural observation scale [McGrath et al,1985]. Pain will be evaluated at arriving in the PACU, 1-hourly during the PACU stay, 4-hourly on the ward, and twice daily after discharge (see questionnaire). Sleeping children will not be woken up.

Cumulative doses per day of paracetamol/codeine and of any other analgesic (NSAIDs, opioids) will be recorded.

Further endpoints

* Quality of sleep during each the night until the surgical visit. Each morning, the care-giver (nurse, parent) will estimate the child's quality of sleep on a NRS ranging from 0=did not sleep at all to 10=excellent sleep.
* First oral intake of fluid (including ice cream); hours after end of surgery.
* First oral intake of solid food; hours after end of surgery.
* At discharge: Overall "satisfaction" judged by the nurse on a NRS ranging from 0=not satisfied at all to 10=very much satisfied.
* Degree of stress on the part of the parents due to the child's "illness". Rated by the parents on a daily basis on a NRS scale from 0=not stressed at all to 10=very much stressed.
* At the surgical visit: Overall "satisfaction" judged by the parents on a NRS ranging from 0=not satisfied at all to 10=very much satisfied.

Adverse effects, safety

* Any minor complication: definition: no need for readmission.
* Any major complication: definition: does need readmission (for instance, readmission due to bleeding, re-operation due to bleeding).

ELIGIBILITY:
Inclusion criteria:

* Elective tonsillectomy with or without adenoidectomy with or without eartubes

Exclusion criteria:

* ASA > II
* Allergie to Dexamethasone
* Recent therapy with steroids or immunotherapy
* Mental retardation
* Children experiencing nausea or vomiting or have taken antiemetic medication within 24 hours before surgery
* Additional surgery
* Enrolement in another investigational study
* Chronic infection or diabetes
* Recent vaccination (less than 1 month prior to surgery)
* Recent varicella infection (less than 1 month prior to surgery)

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Investigation of the dose-effect relationship of prophylactic single-dose dexamethasone for the prevention of postoperative nausea and vomiting in children undergoing adeno-tonsillectomy | 24 hours postoperatively

SECONDARY OUTCOMES:
Dose-effect relationship for the prevention of postoperative pain | 24 hours postoperatively
Oral intake | 10 days
Effect on general outcome | 10 days
Investigation of safety (drug-related harm) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, MBA, Principal Investigator — anesthesia department; Martin Tramer, MD, PhD, Study Chair — anesthesia department
Locations (1):
- University Hospital of Geneva, Anesthesia Department, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Result] Czarnetzki C, Elia N, Lysakowski C, Dumont L, Landis BN, Giger R, Dulguerov P, Desmeules J, Tramer MR. Dexamethasone and risk of nausea and vomiting and postoperative bleeding after tonsillectomy in children: a randomized trial. JAMA. 2008 Dec 10;300(22):2621-30. doi: 10.1001/jama.2008.794. PMID 19066382